CLINICAL TRIAL: NCT05620849
Title: A Technology-based Intervention for Alcohol-related Sexual Risk Behaviors in Young Women
Brief Title: Young Adult Education on Alcohol & Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jessica Blayney, Principal investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010940; 1K99AA028777-01 (NIH); 4R00AA028777 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Sexual Behavior; Alcohol Drinking; Condomless Sex
MeSH Terms: conditions — Sexual Behavior; Alcohol Drinking; Unsafe Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention only (Experimental): This group will complete 4 weeks of the brief online program along with 5 weeks of check-in surveys.
  Interventions: Behavioral: Online program
- Assessment only (No Intervention): This group will complete 5 weeks of check-in surveys.

INTERVENTIONS:
Behavioral: Online program — The online program is 4 weeks and focused on topics such as alcohol and sexual health
  Arms: Intervention only

SUMMARY:
The goal of this clinical trial is to test the effectiveness of our brief online program when compared to those who don't complete the program at all.

DETAILED DESCRIPTION:
A total of 300 participants will complete this 6 month study. The study will include a background survey, 5 week monitoring period where participants either complete the brief online program with check-in surveys or check-in surveys only, and follow-up surveys 1, 3, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Assessed as part of screening procedures

Exclusion Criteria:

* Do not want to participate

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Enrollment is based on female birth sex and female gender identity
Enrollment: 300 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Drinking before sex (frequency) | Follow up (1 month, 3 month, 6 months)
  Using items from the Sexual Health Questionnaire, the investigators will assess the frequency of drinking before sex.
Drinking before sex (quantity) | Follow up (1 month, 3 month, 6 months)
  Using items from the Sexual Health Questionnaire, the investigators will assess the number of drinks consumed before sex.
Condomless sex | Follow up (1 month, 3 month, 6 months)
  Using items from the Sexual Health Questionnaire, the investigators will assess the frequency of condom use during penetrative sex.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Blayney, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No